CLINICAL TRIAL: NCT06623630
Title: A Pilot Safety and Feasibility Study of Lymphodepleting Total Body Irradiation (TBI) Plus Cyclophosphamide Prior to Ciltacabtagene Autoleucel (Carvykti; Cilta-cel) for Multiple Myeloma (MM) Patients With Impaired Renal Function
Brief Title: Lymphodepleting Total Body Irradiation (TBI) Plus Cyclophosphamide Prior to Ciltacabtagene Autoleucel (Carvykti; Cilta-cel) for Multiple Myeloma (MM) Patients With Impaired Renal Function
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Washington University School of Medicine (Other)
Collaborators: American Cancer Society, Inc. (Other); Cures Within Reach (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 202410010
Record Dates: First submitted 2024-09-30; First posted 2024-10-02 (Actual); Last update posted 2025-12-29 (Actual); Status verified 2025-12

CONDITIONS: Multiple Myeloma
Keywords: Chimeric antigen receptor T cells; Radiation; Immunotherapy; Renal failure
MeSH Terms: conditions — Multiple Myeloma; Renal Insufficiency | interventions — Cyclophosphamide; Whole-Body Irradiation

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: Yes | US Export: No

ARMS (1):
- Cyclophosphamide + Cilta-Cel + TBI (Experimental): All patients will undergo T-cell collection and CAR T manufacturing as per standard of care. Patients will receive cyclophosphamide per standard of care Day -5 to Day -3. They will subsequently receive TBI on Day -1 then and will receive cilta-cel infusion on Day 0.
  Interventions: Drug: Cyclophosphamide; Drug: Ciltacabtagene Autoleucel; Radiation: Total body irradiation

INTERVENTIONS:
Drug: Cyclophosphamide — Standard of care
Drug: Ciltacabtagene Autoleucel — Standard of care
  Other Names: Carvykti; cilta-cel
Radiation: Total body irradiation — Radiation doses delivered to the entire body
  Other Names: TBI

SUMMARY:
Treatment for relapsed/refractory multiple myeloma continues to evolve with the approval of highly effective anti-BCMA CAR T therapies in recent years. However, despite the high prevalence of renal insufficiency in this population, pivotal clinical trials have excluded patients with impaired renal function, leading to an urgent, unmet clinical need to develop safe and effective lymphodepleting regimens prior to CAR T administration for this population. In addition, renal insufficiency is linked to poor disease-related outcomes and is highly associated with several underserved populations.

This study is testing the hypotheses that:

1. low-dose total body irradiation (TBI) in combination with cyclophosphamide (Cy) as lymphodepletion prior to administration of cilta-cel will be safe and tolerable in patients with multiple myeloma who have impaired renal function
2. low-dose TBI-Cy as lymphodepletion prior to cilta-cel will result in comparable CAR T expansion/persistence and disease response rates as those seen with standard lymphodepleting chemotherapy (fludarabine / cyclophosphamide).

ELIGIBILITY:
Inclusion Criteria:

* Histologically confirmed diagnosis of multiple myeloma.
* Renal insufficiency, defined as eGFR < 45 by MDRD formula.
* At least 18 years of age.
* ECOG performance status ≤ 1.
* Meets standard of care indication for cilta-cel (per FDA approval).
* Patients with a history of prior autologous hematopoietic cell transplant (AHCT) must have received a graft containing ≥2.0 x 106 CD34+ cells/kg body weight.
* Patients must have adequate cryopreserved autologous stem cells available (≥2.0 x 106 CD34+ cells/kg body weight) in case of prolonged cytopenias to allow for an autologous stem cell boost.
* Women of childbearing potential and men must agree to use adequate contraception prior to study entry and for the duration of study participation. Should a woman become pregnant or suspect she is pregnant while participating in this study or should a man suspect he has fathered a child, s/he must inform her treating physician immediately.
* Ability to understand and willingness to sign an IRB approved written informed consent document. Legally authorized representatives may sign and give informed consent on behalf of study participants.

Exclusion Criteria:

* Prior or concurrent malignancy whose natural history has the potential to interfere with the safety or efficacy assessment of the investigational regimen. Patients with prior or concurrent malignancy that does NOT meet that definition are eligible for this trial.
* Currently receiving any other investigational agents.
* Uncontrolled intercurrent illness including, but not limited to: ongoing or active infection, symptomatic congestive heart failure, unstable angina pectoris, or unstable cardiac arrhythmia. Patients with a known history or current symptoms of cardiac disease, or history of treatment with cardiotoxic agents, should have a clinical risk assessment of cardiac function using the New York Heart Association Function Classification; to be eligible for this trial, patients should be a class 2B or better.
* Pregnant and/or breastfeeding. Women of childbearing potential must have a negative pregnancy test within 14 days of study entry.
* HIV-infected if not on effective anti-retroviral therapy with undetectable viral load for 6 months. Patients with HIV who are receiving effective anti-retroviral therapy and have had an undetectable viral load for at least 6 months are eligible.
* Evidence of chronic hepatitis B virus (HBV) that is detectable on suppressive therapy. Patients with evidence of chronic HBV infection with undetectable HBV viral load on suppressive therapy are eligible.
* History of hepatitis C virus (HCV) infection that has not been cured or that has a detectable viral load. Patients with a history of HCV that has been treated and cured are eligible. Patients with HCV infection who are currently on treatment and have an undetectable HCV viral load are eligible.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 12 (Estimated)
Dates: Start 2024-12-04 (Actual); Primary Completion 2026-04-30 (Estimated); Study Completion 2027-03-31 (Estimated)

PRIMARY OUTCOMES:
Incidence of dose-limiting toxicities (DLTs) | Through 28 days post cilta-cel
  Toxicities considered possibly, probably, or definitely related to TBI-based lymphodepletion as graded per CTCAE v 5.0.

SECONDARY OUTCOMES:
Incidence of treatment related adverse events (TEAEs) | Through completion of follow-up (estimated to 1 year and 1 week)
  * Graded per CTCAE v 5.0.
  * All AEs will be collected from start of treatment through Day 28. After Day 28, only late toxicities of interest will be tracked and recorded.
Incidence of cytokine release syndrome (CRS) | Through day 100
Incidence of immune effector cell associated neurotoxicity syndrome (ICANS) | Through day 100
  Graded per ASTCT criteria
Best overall response by IMWG criteria | Through completion of follow-up (estimated to 1 year and 1 week)
Response rate by IMWG criteria | Day 28 post cilta-cel
Response rate by IMWG criteria | Day 100 post cilta-cel
Response rate by IMWG criteria | 1 year post cilta-cel
Measurable residual disease (MRD) as measured by ClonoSeq | Day 28 post cilta-cel
Measurable residual disease (MRD) as measured by ClonoSeq | Day 100 post cilta-cel
Measurable residual disease (MRD) as measured by ClonoSeq | 1 year post cilta-cel
Median duration of response (DoR) | Through completion of follow-up (estimated to 1 year and 1 week)
  Duration of response (DoR) is defined as the time from onset of response to progression or death due to any reason, whichever occurs earlier.
Duration of response | Through completion of follow-up (estimated to 1 year and 1 week)
  Duration of response (DoR) is defined as the time from onset of response to progression or death due to any reason, whichever occurs earlier.
Progression-free survival (PFS) | Through completion of follow-up (estimated to 1 year and 1 week)
  Progression-free survival (PFS) is defined as the time from start of treatment (Day 0) until date of disease progression.
Overall survival (OS) | Through completion of follow-up (estimated to 1 year and 1 week)
  Overall survival (OS) is defined as the time from start of treatment (Day 0) until date of death.
Area under the curve (AUC) for CAR T expansion as measured by multiparameter flow cytometry. | Through completion of follow-up (estimated to 1 year and 1 week)
Area under the curve (AUC) for CAR T expansion as measured by quantitative polymerase chain reaction (qPCR). | Through completion of follow-up (estimated to 1 year and 1 week)

CONTACTS AND LOCATIONS:
Overall Officials: Michael J Slade, M.D., MSCI, Principal Investigator — Washington University School of Medicine
Locations (1):
- Washington University School of Medicine, St Louis, Missouri, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: Alvin J. Siteman Cancer Center at Barnes-Jewish Hospital and Washington University School of Medicine — http://www.siteman.wustl.edu